CLINICAL TRIAL: NCT05591625
Title: A Multi-centre, Randomised, Pilot Feasibility Study to Compare the Effectiveness of Eye-movement Desensitisation and Reprocessing Versus Usual Care in the Psychological Recovery of Intensive Care Survivors
Brief Title: Eye Movement Desensitisation and Reprocessing (EMDR) to Improve Mental Health Following Intensive Care Admission
Acronym: EMERALD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHM CRI0424
Record Dates: First submitted 2022-10-06; First posted 2022-10-24 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Post Traumatic Stress Disorder; Critical Illness; Eye Movement Desensitisation and Reprocessing; Depression, Anxiety
Keywords: EMDR; Feasibility; Acceptability
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Critical Illness; Depression; Anxiety Disorders | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: Participants with PTSD symptoms (2-3 months post-hospital discharge) will be assigned to either usual care or usual care plus EMDR.
  Participants without PTSD symptoms (2-3 months post-hospital discharge) will enter an observation arm, which consists of a repeat psychological assessment at 12-months post-hospital discharge.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants who exhibit symptoms of PTSD and are randomised to the control group, will receive usual care offered by their hospital.
- Eye Movement Desensitisation and Reprocessing (Experimental): Participants who exhibit symptoms of PTSD and are randomised to the intervention group, will receive EMDR plus usual care offered by their hospital. EMDR will be delivered by trained and accredited psychological therapists, employed by National Health Service community mental health teams.
  Interventions: Behavioral: Eye Movement Desensitisation and Reprocessing
- Observation (No Intervention): Participants who do not exhibit symptoms of PTSD will receive usual care offered by their hospital and repeat the psychological assessment at 12-months post-hospital discharge.

INTERVENTIONS:
Behavioral: Eye Movement Desensitisation and Reprocessing — EMDR is a trauma-focussed, psychological talking therapy whereby the participant verbally relates a narrative of an emotionally disturbing memory, in brief sequential doses, while simultaneously focusing on an external stimulus, most commonly side-to-side finger movements of the psychological therapist. EMDR aims to enable an individual to process memories of the event in order to reduce psychological morbidity. EMDR is widely practiced, so is scalable. It is also protocolised, so can be taught and tested, and allows for fidelity assessment in controlled studies.
  The number of sessions will depend on ongoing presence of disturbing memories. This will be determined by the psychological therapist and participant.
  Other Names: EMDR
  Arms: Eye Movement Desensitisation and Reprocessing

SUMMARY:
The goal of this multi-centre, randomised, pilot feasibility study is to assess the feasibility of recruiting intensive care survivors, with symptoms of traumatic stress, to a study evaluating the use of eye movement desensitisation and reprocessing (EMDR). The main purpose is to determine whether it is feasible and acceptable to patients, clinicians and researchers. In addition, this study aims to identify design criteria that may be of use in a subsequent randomised controlled trial of clinical effectiveness.

Participants will:

* be recruited at hospital discharge
* undergo a psychological assessment at 2-3 months post-hospital discharge
* Those exhibiting symptoms of post-traumatic stress disorder (PTSD), will be randomised (1:1) to receive either usual care or usual care plus EMDR
* Participants who do not exhibit PTSD symptoms at the 2-3 month assessment will enter a light-touch observation arm.
* All participants will repeat the psychological assessment 12-months after hospital discharge.

Feasibility parameters; recruitment, adherence, retention and safety data. Primary clinical outcomes; change in PTSD symptoms between 2-3 months and 12-months.

The investigators will undertake a qualitative process evaluation using clinical ethnography and reported according to the Theoretical Framework of Acceptability.

DETAILED DESCRIPTION:
Background:

Patients who survive a period of critical illness have a disproportionately high chance of suffering from disturbing and persistent downstream psychological morbidity. These are associated with reduced quality of life and increased healthcare utilisation.

A recent survey of United Kingdom follow-up services reported a lack of post-discharge psychological support. There have been calls for collaborative efforts, between ICU and mental health professionals, exploring whether established trauma-focussed treatment modalities, may be tested for the benefit of ICU survivors.

Eye-Movement Desensitisation and Reprocessing (EMDR) has improved mental health in combat veterans and victims of man-made and natural disasters. Small studies have also shown it to be effective in healthcare settings, within the Emergency department, following cancer diagnosis and implantation of cardioverter defibrillators. EMDR is recommended by United Kingdom National Institute for Health and Care Excellence, World Health Organisation and the Institute for Traumatic Stress Studies, for treating adult onset PTSD.

The investigators hypothesise that post-intensive care psychological health will be improved by EMDR. Reports of it's application in this cohort have largely adopted a case study approach. EMDR has never been systematically evaluated for effect in intensive care survivors.

The investigator's recently completed feasibility study (NCT04455360) (In press; Journal of the Intensive Care Society) informed design refinements for this study. Prior to conducting a large scale study of clinical effectiveness, it is important to answer remaining uncertainties, regarding feasibility, acceptability and to identify potential adaptations to trial design.

Aims:

* To evaluate whether it is feasible and acceptable to investigate EMDR, for intensive care survivors in a clinical trial.
* To inform refinements to the design of a fully-powered randomised controlled trial (RCT) of clinical effectiveness.
* To determine preliminary clinical effect of EMDR on PTSD symptoms of traumatised survivors of intensive care admission.

Method:

A mixed methods, multi-centre, fully-randomised controlled, patient preference, pilot feasibility study.

Patients will be recruited from University Hospital Southampton ICU, Royal Bournemouth Hospital ICU, Poole General Hospital ICU and Queen Alexandra Hospital ICU, Portsmouth in the United Kingdom.

All participants will enter a common pathway, watch and wait study, between Part A consent and the 2-month post-hospital discharge assessment.

Part A: Watch and wait consent Hospital research staff will screen all patients within the ICU. Patients who fulfil inclusion criteria but have none of the exclusion criteria will be approached to discuss trial participation. The patient will be given the Patient Information Sheet (PIS) and adequate time to consider participation according to Good Clinical Practice guidelines. Capacity to consent must be determined in accordance to the Mental Capacity Act 2005.

Two month psychometric assessment All participants who granted Part A consent, to the 'watch and wait' study will be invited to undertake screening for PTSD symptoms using the Impact of Events Scale-Revised (IES-R). This patient-rated outcome measure can be completed electronically by following a link sent via email. Alternatively, paper versions can be posted, with a stamped addressed return envelope included.

Participants with a total IES-R score ≥22, indicative of symptoms of post-traumatic stress, will be invited to consider consenting to an RCT of EMDR vs usual care.

Non-symptomatic participants (IES-R≤21) and those who are unwilling or unable to participate in the RCT, will be asked to continue in the observation study, by completing the 12-month psychometric assessment.

Part B: RCT consent The study team will telephone participants, who score ≥22 on the 2-month PTSD screen, and ask them to consider consenting to the RCT of EMDR vs usual care. The RCT participant information sheet (PIS) and informed consent form (ICF) will be available electronically or via post. Participants consenting to the RCT will be asked to undertake a Clinical Administered PTSD Scale for Diagnostic Statistical Manual-5 (CAPS-5) assessment of PTSD symptoms and a Clinical Global Impression of Illness Severity (CGI-S). In addition, the research team will ask participants to rate which arm of the study they would prefer, using a Likert scale of 0-10.

Following this assessment, the study team will ask participants, with symptoms of post-traumatic stress, to consider entering an RCT of EMDR vs usual care. (Part B consent) Participants who are not displaying symptoms of post-traumatic stress will be asked to enter an observation arm, and repeat the assessment, 12-months post-hospital discharge.

Participants who consent to Part B of the study will be randomised 1:1 to either usual care or usual care plus EMDR with their local National health Service Psychological service.

All participants will repeat the 12-month assessment.

The investigators will conduct a qualitative process evaluation to capture contextual and cultural factors not adequately determined by a purely quantitative study.

If feasibility and acceptability are established, information from this study will inform the design of a subsequent, fully-powered Randomised Controlled Trial, to determine whether EMDR is an effective treatment option for post-intensive care psychological health.

ELIGIBILITY:
Inclusion Criteria:

* Survivors of an intensive care admission, who have received level 3 care for >24 hours.
* Aged ≥18 years
* Capacity to provide informed consent and complete trial interventions and assessments.

Exclusion Criteria:

* Pre-existing cognitive impairment such as dementia
* Pre-existing diagnosis of psychosis
* Not expected to survive post-hospital discharge
* Traumatic brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Recruitment, adherence, retention | 12-months
  To determine whether investigating the use of EMDR for traumatised survivors of critical care can reach predefined feasibility objectives:
  * Recruitment rate part A - we anticipate an average recruitment of 10 patients per month across the three participating sites. This is well above the median recruitment of 0.95 participants recruited per site per month, reported in a review of trials listed in the NIHR journals library (1997-2020)(31).
  * Consent rate - number of patients recruited, expressed as a percentage of patients approached. Based on our previous work we expect this to be greater than 30%(28).
  * Adherence will be determined by completion of ≥75% of planned EMDR sessions completed.
  * Retention will be determined by ≥75% of participants completing the study follow-up assessment.
Acceptability | 12-months
  To explore acceptability of participating in a Randomised Controlled Trail of EMDR for critical care survivors, psychology clinicians and research staff. Reported according to the Theoretical Framework of Acceptability. This qualitative methodology, using semi-structured interviews, provides a framework for assessing conceptually different constructs of acceptability in clinical trials; affective attitude, burden, ethicality, intervention coherence, opportunity costs, perceived effectiveness and self-efficacy.
Number of participants with adverse events (safety and tolerability) | 12-months
  Safety will be determined by assignment of causality of serious events. Events attributable to trial procedures will be reviewed by trial management board, study sponsor and the research ethics committee, in order to determine ongoing feasibility.

SECONDARY OUTCOMES:
Post-traumatic stress disorder | 12-months
  Change in post-traumatic stress disorder (PTSD) symptom severity using the Impact of Events Scale-Revised. (IES-R) The IES-R is a 22-question, patient reported outcome measure widely used to assess symptoms of PTSD, including in critical care research, and is recommended by critical care core outcome dataset developers and the International Conference of Harmonisation of Outcome Measures. The questions cover symptoms of intrusion, avoidance and hyperarousal. Participants indicate how distressing the symptoms have been over the last 7 days. Symptom severity can be 0 (not at all), 1 (a little bit), 2 (moderately), 3 (quite a bit), 4 (extremely), giving a total scoring range of 0 to 88, with higher scores indicating more severe symptoms.
Clinician assessed Post-traumatic stress disorder | 12-months
  To determine changes in symptoms of PTSD, participants will undergo the Clinician administered PTSD scale (CAPS-5) assessment at 2- and 12-months post-hospital discharge.
  CAPS-5 is a 30-question structured interview, exploring severity and duration of PTSD symptoms, index trauma, subjective distress and impact on social and occupational functioning. Each question refers to PTSD symptoms and can be rated; 0=absent; 1=mild/sub-threshold; 2=moderate/threshold; 3=severe/markedly elevated; 4=extreme/incapacitating.
  Scores from questions 1-20 will be combined to give an overall severity ranging, with high scores reflecting worse symptoms. In addition, the investigators will sum individual symptoms relating to symptom clusters from the Diagnostic and Statistical Manual of mental disorder; (5th Ed)
Sensitivity analysis | 12-months
  To determine whether PTSD symptom severity and diagnoses, identified by patent reported Impact of Events Scale-Revised, correspond with those identified by Clinician administered PTSD Scale-5.
Anxiety | 12-months
  Generalised Anxiety Disorder-7 (GAD-7): this 7-question, self-administered tool is validated to assess for anxiety symptom severity. Scores are calculated by assigning 0 for 'not at all, 1- 'several days', 2 - 'more than half the days' or 3 - 'nearly every day' for responses to nine questions, giving a score in the range 0-21. GAD-7 scores of 5, 10 and 15 represent cut-offs for mild, moderate and severe anxiety respectively.
Depression | 12-months
  Patient Health Questionnaire-9 (PHQ-9): this self-administered, validated tool assesses depressive symptom severity. Scores are calculated by assigning 0 for 'not at all, 1- 'several days', 2 - 'more than half the days' or 3 - 'nearly every day' for responses to nine questions, giving a score in the range 0-27. PHQ-9 score of 0-4 demonstrates no - minimal depression severity. 5-9 = mild severity, 10-14 = moderate severity, 15-19 = moderately severe, 20-27 = severe.
Health related quality of life | 12-months
  EuroQol Five Dimension- Five level scale (EQ5D -5L): comprises five quality-of-life dimensions; mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Participants report levels ranging from 'no problems' to 'extreme problems'.
Clinical Global Impression of Improvement (CGI-I) | 12-months
  The Clinical Global Impression of improvement can be used to assess symptom severity and response to treatment. It requires a clinician to rate the severity of a patient's mental illness, relative to other patients that the clinician has seen, who have the same diagnosis. The 7-point scale ranges from; 1 - normal, not at all ill, 2 - borderline mentally ill, 3 - mildly ill, 4 - moderately ill, 5 - markedly ill, 6 - severely ill, 7 - among the most extremely ill patients.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University Hospitals Dorset, Poole, Dorset
  - University Hospital Southampton, Southampton, Hampshire

IPD SHARING:
Plan to Share IPD: No
Researchers should contact the Chief Investigator. The decision to share Individual Participant Data will be determined on a case-by-case basis.

REFERENCES:
- [Derived] Bates A, Golding H, Rushbrook S, Highfield J, Pattison N, Baldwin D, Grocott MPW, Cusack R. Mixed-methods randomised study exploring the feasibility and acceptability of eye-movement desensitisation and reprocessing for improving the mental health of traumatised survivors of intensive care following hospital discharge: protocol. BMJ Open. 2024 Jan 29;14(1):e081969. doi: 10.1136/bmjopen-2023-081969. PMID 38286705